CLINICAL TRIAL: NCT01497054
Title: Diagnostic Prediction Value of B Type Natriuretic Peptide (BNP) Levels in Hemodynamically Significant Patent Ductus Arteriosus (hsPDA) in Premature Infants.
Brief Title: Do Elevated BNP Levels Predict Hemodynamically Significant PDAs
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Collaborators: Alere, Inc. (Industry)
Responsible Party: Principal Investigator, Kate Tauber, Principal Investigator, Albany Medical College
Other Study IDs: 3155
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2011-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: B type natriuretic peptide; Patent Ductus Arteriosus; Preterm infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if B type natriuretic peptide (BNP) levels can be used to predict a hemodynamically significant patent ductus arteriosus (PDA). This peptide is produced by the ventricles in the heart when they are under stress, such as when a ductus remains open. If we can use a simple and inexpensive blood test to determine whether a PDA needs to be treated, we can potentially treat infants sooner than if they needed to wait for the availability of a cardiologist to perform an echocardiogram. This might decrease some of the deleterious effects of PDAs on the preterm infant such as bronchopulmonary dysplasia, necrotizing enterocolitis, renal hypoperfusion, and pulmonary hemorrhage. In a situation where follow up echocardiogram after a course of medical therapy shows persistent PDA, this test may help to decide whether this baby needs further treatment, either medical or surgical.

DETAILED DESCRIPTION:
B type natriuretic peptide (BNP) is mainly synthesized in the ventricles of the heart and released in response to volume and pressure loading and ventricular stress and, therefore, plays an important role in regulation of extracellular fluid volume. BNP causes diuresis, natriuresis, arterial and venous vasodilation and antagonizes the renin-angiotensin system resulting in a reduction in intravascular volume and decreased ventricular preload and afterload.

In adults, BNP levels have been routinely used to diagnose and measure the degree of congestive heart failure. In healthy term infants, BNP levels are initially elevated in the first few days of life but then decline over the ensuing week after birth to near adult levels by 3 months of age. However, in premature newborn infants there are still no normative values for BNP and, therefore, no agreed-upon cut off points to diagnose ventricular overload without confirmatory echocardiography. Patent ductus arteriosus (PDA) is the most common cause of ventricular overload and congestive heart failure in premature neonates and can be a cause of significant morbidity. Excessive pulmonary blood flow due to the aortopulmonary shunting can result in increased ventilatory dependency and thereby contribute to chronic lung disease. Other possible sequelae from a PDA include renal hypoperfusion, necrotizing entercolitis, and pulmonary hemorrhage. Early closure of a PDA has been shown to reduce these risks.

Delayed ductal closure is inversely related to GA at birth with the incidence varying from 20% in babies greater than 32 weeks gestation and up to 60% in babies less than 28 weeks gestation. Currently, infants are screened for a PDA by echocardiography. This requires that centers have access to cardiologists to perform and analyze these studies. A simple blood test that could help diagnose a hemodynamically significant PDA would be extremely helpful in low birth weight infants, especially in more remote centers that do not have routine access to cardiology services. To date, there is no accepted blood test although numerous studies are emerging suggesting that BNP might be such a test. It has been shown that the magnitude of shunting through a PDA is a major determinant of BNP level, however, the levels published in various studies for what is hemodynamically significant varies greatly. In addition, the studies that have been done previously are on small sample sizes (less than 70 patients, with one retrospective study that had 88 patients) and on various gestational ages and, therefore, it is difficult to extrapolate normative data.

It is already known that BNP levels are elevated in neonates with a hsPDA, however, there is little agreement on how high a BNP level needs to get to imply a hsPDA. We propose a study to measure the BNP values in all infants born less than 32 weeks gestation with and without a PDA. We will also do serial BNP levels with concurrent echocardiograms in infants with a PDA to determine a cutoff value of BNP above which an infant is likely to have a hsPDA. We hope that our study, with a larger sample size and on all infants with and without a PDA, will be able to not only gather more definitive data on what the cutoff BNP level is, but also gather normative BNP data on premature infants without PDAs.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 24 0/7 weeks gestation and 31 6/7 weeks gestation. - Infants must be enrolled by 24 hours of life.

Exclusion Criteria:

* congenital heart disease,
* necrotizing enterocolitis,
* culture positive sepsis or culture negative but treated for presumed sepsis.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants between 24 0/7 weeks gestation and 31 6/7 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
BNP level and size of PDA | within first 2 weeks of life
  BNP levels measured at several time points during first 2 weeks of life and compared to findings on echocardiogram to see if size of PDA correlated with BNP level.

CONTACTS AND LOCATIONS:
Overall Officials: Kate A Tauber, MD, Principal Investigator — Albany Medical College; Upender K Munshi, MD, Study Director — Albany Medical College; Robin Doyle, MD, Study Director — Capital Distric Pediatric Cardiology, affiliated with Albany Medical Center
Locations (1):
- Albany Medical Center Neonatal Intesive Care Unit, Albany, New York, United States

REFERENCES:
- [Background] Sanjeev S, Pettersen M, Lua J, Thomas R, Shankaran S, L'Ecuyer T. Role of plasma B-type natriuretic peptide in screening for hemodynamically significant patent ductus arteriosus in preterm neonates. J Perinatol. 2005 Nov;25(11):709-13. doi: 10.1038/sj.jp.7211383. PMID 16222347
- [Background] Holmstrom H, Hall C, Thaulow E. Plasma levels of natriuretic peptides and hemodynamic assessment of patent ductus arteriosus in preterm infants. Acta Paediatr. 2001 Feb;90(2):184-91. doi: 10.1080/080352501300049406. PMID 11236049